CLINICAL TRIAL: NCT00647374
Title: Assessment of Cortical Plasticity Following Short Term Limb Immobility
Status: Suspended | Type: Observational
Sponsor: Hadassah Medical Organization (Other)
Other Study IDs: NETTA001-HMO-CTIL
Record Dates: First submitted 2008-03-26; First posted 2008-03-31 (Estimated); Last update posted 2010-03-02 (Estimated); Status verified 2010-02

CONDITIONS: Fracture
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- 1
  Interventions: Other: this is an observational study

INTERVENTIONS:
Other: this is an observational study

SUMMARY:
The proposed project will study the consequence of short term limb immobility on the patterns of brain activity using functional imaging (fMRI)

ELIGIBILITY:
Inclusion Criteria:

* wrist fracture.
* Fit for MRI scanning.

Exclusion Criteria:

* Unwillingness to sign informed consent.
* Neurological disease
* s/p fractures

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with wristfracture
Sampling Method: Non-Probability Sample
Dates: Start 2008-05

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization., Jerusalem, Israel